CLINICAL TRIAL: NCT04909671
Title: Evaluation of ArTificial Intelligence System (Gi-Genius) for adenoMa dEtection in Lynch Syndrome. A Randomized, Parallel, Multicenter, Controlled Trial. TIMELY Study.
Brief Title: Evaluation of ArTificial Intelligence System (Gi-Genius) for adenoMa dEtection in Lynch Syndrome.
Acronym: Timely
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: European Society of Gastrointestinal Endoscopy (Other)
Responsible Party: Principal Investigator, María Pellisé, Principal Investigator. Attending physician Gastroenterology department., Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: Timely
Record Dates: First submitted 2021-05-21; First posted 2021-06-02 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Lynch Syndrome
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAD arm (Active Comparator): Patients allocated to CAD arm will receive during colonoscopy withdrawal high definition white light endoscopy aided with artificial intelligence device (Gi Genius, Medtronic)
  Interventions: Device: Gi Genius, Medtronic
- WLE arm (Placebo Comparator): Patients allocated to WLE arm will receive during colonoscopy withdrawal high definition white light endoscopy as standart of care.
  Interventions: Other: White light standart colonoscopy

INTERVENTIONS:
Device: Gi Genius, Medtronic — GI geniusTM (Medtronic) is an artificial intelligence device designed and validated on a dataset of white-light endoscopy videos from high-quality randomized controlled trials for the detection of colorectal lesions during colonoscopy. Based on a deep learning system using convolutional neural networks, GI genius works in real-time side-to-side with the gastroenterologist during colonoscopy highlighting the presence of precancerous lesions with a visual marker (green box) in real time and designed to be integrated with the majority of colonoscopies.
  Arms: CAD arm
Other: White light standart colonoscopy — High definition white light endoscopy will be used during the scope withdrawal
  Arms: WLE arm

SUMMARY:
The purpose of this study is to assess if artificial intelligence aid colonoscopy colonoscopy is superior to conventional colonoscopy for the detection of adenomas during surveillance colonoscopy in patients with Lynch syndrome.

DETAILED DESCRIPTION:
To compare the performance of white-light colonoscopy (HD-WLE) versus white-light + CAD (CAD) for detection of adenomas (1:1 ratio). The CAD system will include an artificial intelligence-based medical device (GI Genius, Medtronic) trained to process colonoscopy images and superimpose them, in real time, on the endoscopy display as a green box over suspected lesion. An adequate bowel preparation and minimum withdrawal time of 6 min will be required. Colonoscopies will be performed by experienced endoscopists and with high-definition scopes. Lesions will be collected, and histopathology findings used as the reference standard. The primary outcome of this trial will be the mean number of adenomas per colonoscopy (APC).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years with a proven pathogenic germline variant in one of the MMR genes (MLH1, MSH2, MSH6) or Epcam deletion who are under surveillance colonoscopy.

Exclusion Criteria:

* Previous history of total colectomy,
* Concomitant inflammatory bowel disease,
* Inability or refuse to sign the informed consent,
* Previous colonoscopy < 12 months.
* Inadequate bowel preparation.
* Incomplete procedure.
* PMS2 mutation carriers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Estimated)
Dates: Start 2021-09-13 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Mean number of adenomas per colonoscopy | 18 months
  Compare mean number of adenomas in both arms calculated by dividing the total number of adenomas detected by the total number of colonoscopies in each arm

SECONDARY OUTCOMES:
Withdrawal time | 18 months
  time spent on inspection, from the cecum to endoscope extraction through the anus, excluding the time needed for therapeutic measures (including polypectomy).
Mean number of polyps per colonoscopy | 18 months
  Compare mean number of polyps in both arms calculated by dividing the total number of polyps (including serrated lesions and adenomas) detected by the total number of colonoscopies in each arm
Adenoma detection rate | 18 months
  proportion of individuals undergoing a complete colonoscopy who had at least one adenoma detected between two arms.
Polyp detection rate | 18 months
  proportion of individuals undergoing a complete colonoscopy who had at least one polyp detected between two arms.
False positives in CAD arm | 18 months
  Combination of:
  * Lesions detected by CAD (>2s green box) after an adequate inspection with a high confidence optical diagnosis negative for neoplasia made by the endoscopist.
  * Lesions detected by CAD (>2s green box) after an adequate inspection resected by the endoscopist and with a clinically non-significant histology.
Mean number of non-clinically significant removed lesions | 18 months
  Lesions removed and with a histology of normal or inflammatory mucosa or removed diminutive recto-sigmoid polyps with a histology of hyperplastic
Subjective endoscopist measures | 18 months
  Questionary addresing the easiness and satisfaction of the procedure, detection of lesions and performance of artificial intelligence will be filled in by each endoscopist

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - María Pellisé. MD. PhD., Barcelona
  - Oswaldo ortiz, Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lynch HT, Snyder CL, Shaw TG, Heinen CD, Hitchins MP. Milestones of Lynch syndrome: 1895-2015. Nat Rev Cancer. 2015 Mar;15(3):181-94. doi: 10.1038/nrc3878. Epub 2015 Feb 12. PMID 25673086
- [Background] Haraldsdottir S, Rafnar T, Frankel WL, Einarsdottir S, Sigurdsson A, Hampel H, Snaebjornsson P, Masson G, Weng D, Arngrimsson R, Kehr B, Yilmaz A, Haraldsson S, Sulem P, Stefansson T, Shields PG, Sigurdsson F, Bekaii-Saab T, Moller PH, Steinarsdottir M, Alexiusdottir K, Hitchins M, Pritchard CC, de la Chapelle A, Jonasson JG, Goldberg RM, Stefansson K. Comprehensive population-wide analysis of Lynch syndrome in Iceland reveals founder mutations in MSH6 and PMS2. Nat Commun. 2017 May 3;8:14755. doi: 10.1038/ncomms14755. PMID 28466842
- [Background] de Jong AE, Hendriks YM, Kleibeuker JH, de Boer SY, Cats A, Griffioen G, Nagengast FM, Nelis FG, Rookus MA, Vasen HF. Decrease in mortality in Lynch syndrome families because of surveillance. Gastroenterology. 2006 Mar;130(3):665-71. doi: 10.1053/j.gastro.2005.11.032. PMID 16530507
- [Background] Jarvinen HJ, Aarnio M, Mustonen H, Aktan-Collan K, Aaltonen LA, Peltomaki P, De La Chapelle A, Mecklin JP. Controlled 15-year trial on screening for colorectal cancer in families with hereditary nonpolyposis colorectal cancer. Gastroenterology. 2000 May;118(5):829-34. doi: 10.1016/s0016-5085(00)70168-5. PMID 10784581
- [Background] Huneburg R, Lammert F, Rabe C, Rahner N, Kahl P, Buttner R, Propping P, Sauerbruch T, Lamberti C. Chromocolonoscopy detects more adenomas than white light colonoscopy or narrow band imaging colonoscopy in hereditary nonpolyposis colorectal cancer screening. Endoscopy. 2009 Apr;41(4):316-22. doi: 10.1055/s-0028-1119628. Epub 2009 Apr 1. PMID 19340735
- [Background] Rahmi G, Lecomte T, Malka D, Maniere T, Le Rhun M, Guimbaud R, Lapalus MG, Le Sidaner A, Moussata D, Caron O, Barbieux JP, Gaudric M, Coron E, Barange K, Ponchon T, Sautereau D, Samaha E, Saurin JC, Chaussade S, Laurent-Puig P, Chatellier G, Cellier C. Impact of chromoscopy on adenoma detection in patients with Lynch syndrome: a prospective, multicenter, blinded, tandem colonoscopy study. Am J Gastroenterol. 2015 Feb;110(2):288-98. doi: 10.1038/ajg.2014.423. Epub 2015 Jan 20. PMID 25601014
- [Background] East JE, Suzuki N, Stavrinidis M, Guenther T, Thomas HJ, Saunders BP. Narrow band imaging for colonoscopic surveillance in hereditary non-polyposis colorectal cancer. Gut. 2008 Jan;57(1):65-70. doi: 10.1136/gut.2007.128926. Epub 2007 Aug 6. PMID 17682000
- [Background] Rijcken FE, Hollema H, Kleibeuker JH. Proximal adenomas in hereditary non-polyposis colorectal cancer are prone to rapid malignant transformation. Gut. 2002 Mar;50(3):382-6. doi: 10.1136/gut.50.3.382. PMID 11839719
- [Background] De Jong AE, Morreau H, Van Puijenbroek M, Eilers PH, Wijnen J, Nagengast FM, Griffioen G, Cats A, Menko FH, Kleibeuker JH, Vasen HF. The role of mismatch repair gene defects in the development of adenomas in patients with HNPCC. Gastroenterology. 2004 Jan;126(1):42-8. doi: 10.1053/j.gastro.2003.10.043. PMID 14699485
- [Background] Rondagh EJ, Gulikers S, Gomez-Garcia EB, Vanlingen Y, Detisch Y, Winkens B, Vasen HF, Masclee AA, Sanduleanu S. Nonpolypoid colorectal neoplasms: a challenge in endoscopic surveillance of patients with Lynch syndrome. Endoscopy. 2013;45(4):257-64. doi: 10.1055/s-0032-1326195. Epub 2013 Feb 25. PMID 23440588
- [Background] van Leerdam ME, Roos VH, van Hooft JE, Balaguer F, Dekker E, Kaminski MF, Latchford A, Neumann H, Ricciardiello L, Rupinska M, Saurin JC, Tanis PJ, Wagner A, Jover R, Pellise M. Endoscopic management of Lynch syndrome and of familial risk of colorectal cancer: European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2019 Nov;51(11):1082-1093. doi: 10.1055/a-1016-4977. Epub 2019 Oct 9. PMID 31597170
- [Background] Sanchez A, Roos VH, Navarro M, Pineda M, Caballol B, Moreno L, Carballal S, Rodriguez-Alonso L, Ramon Y Cajal T, Llort G, Pinol V, Lopez-Fernandez A, Salces I, Pico MD, Rivas L, Bujanda L, Garzon M, Pizarro A, Martinez de Castro E, Lopez-Arias MJ, Poves C, Garau C, Rodriguez-Alcalde D, Herraiz M, Alvarez-Urrutia C, Dacal A, Carrillo-Palau M, Cid L, Ponce M, Barreiro-Alonso E, Saperas E, Aguirre E, Romero C, Bastiaansen B, Gonzalez-Acosta M, Morales-Romero B, Ocana T, Rivero-Sanchez L, Jung G, Bessa X, Cubiella J, Jover R, Rodriguez-Moranta F, Balmana J, Brunet J, Castells A, Dekker E, Capella G, Serra-Burriel M, Moreira L, Pellise M, Balaguer F. Quality of Colonoscopy Is Associated With Adenoma Detection and Postcolonoscopy Colorectal Cancer Prevention in Lynch Syndrome. Clin Gastroenterol Hepatol. 2022 Mar;20(3):611-621.e9. doi: 10.1016/j.cgh.2020.11.002. Epub 2020 Nov 3. PMID 33157315
- [Background] Rivero-Sanchez L, Arnau-Collell C, Herrero J, Remedios D, Cubiella J, Garcia-Cougil M, Alvarez V, Albeniz E, Calvo P, Gordillo J, Puig I, Lopez-Vicente J, Huerta A, Lopez-Ceron M, Salces I, Penas B, Parejo S, Rodriguez de Santiago E, Herraiz M, Carretero C, Gimeno-Garcia AZ, Saperas E, Alvarez-Urturi C, Moreira R, Rodriguez de Miguel C, Ocana T, Moreira L, Carballal S, Sanchez A, Jung G, Castells A, Llach J, Balaguer F, Pellise M; EndoCAR group from Spanish Gastroenterology Association (AEG) and Spanish Society of Digestive Endoscopy (SEED). White-Light Endoscopy Is Adequate for Lynch Syndrome Surveillance in a Randomized and Noninferiority Study. Gastroenterology. 2020 Mar;158(4):895-904.e1. doi: 10.1053/j.gastro.2019.09.003. Epub 2019 Sep 12. PMID 31520613
- [Background] Repici A, Badalamenti M, Maselli R, Correale L, Radaelli F, Rondonotti E, Ferrara E, Spadaccini M, Alkandari A, Fugazza A, Anderloni A, Galtieri PA, Pellegatta G, Carrara S, Di Leo M, Craviotto V, Lamonaca L, Lorenzetti R, Andrealli A, Antonelli G, Wallace M, Sharma P, Rosch T, Hassan C. Efficacy of Real-Time Computer-Aided Detection of Colorectal Neoplasia in a Randomized Trial. Gastroenterology. 2020 Aug;159(2):512-520.e7. doi: 10.1053/j.gastro.2020.04.062. Epub 2020 May 1. PMID 32371116
- [Background] Hassan C, Spadaccini M, Iannone A, Maselli R, Jovani M, Chandrasekar VT, Antonelli G, Yu H, Areia M, Dinis-Ribeiro M, Bhandari P, Sharma P, Rex DK, Rosch T, Wallace M, Repici A. Performance of artificial intelligence in colonoscopy for adenoma and polyp detection: a systematic review and meta-analysis. Gastrointest Endosc. 2021 Jan;93(1):77-85.e6. doi: 10.1016/j.gie.2020.06.059. Epub 2020 Jun 26. PMID 32598963
- [Background] Endoscopic Classification Review Group. Update on the paris classification of superficial neoplastic lesions in the digestive tract. Endoscopy. 2005 Jun;37(6):570-8. doi: 10.1055/s-2005-861352. PMID 15933932
- [Background] Kaminski MF, Thomas-Gibson S, Bugajski M, Bretthauer M, Rees CJ, Dekker E, Hoff G, Jover R, Suchanek S, Ferlitsch M, Anderson J, Roesch T, Hultcranz R, Racz I, Kuipers EJ, Garborg K, East JE, Rupinski M, Seip B, Bennett C, Senore C, Minozzi S, Bisschops R, Domagk D, Valori R, Spada C, Hassan C, Dinis-Ribeiro M, Rutter MD. Performance measures for lower gastrointestinal endoscopy: a European Society of Gastrointestinal Endoscopy (ESGE) Quality Improvement Initiative. Endoscopy. 2017 Apr;49(4):378-397. doi: 10.1055/s-0043-103411. Epub 2017 Mar 7. PMID 28268235
- [Background] IJspeert JE, Bastiaansen BA, van Leerdam ME, Meijer GA, van Eeden S, Sanduleanu S, Schoon EJ, Bisseling TM, Spaander MC, van Lelyveld N, Bargeman M, Wang J, Dekker E; Dutch Workgroup serrAted polypS & Polyposis (WASP). Development and validation of the WASP classification system for optical diagnosis of adenomas, hyperplastic polyps and sessile serrated adenomas/polyps. Gut. 2016 Jun;65(6):963-70. doi: 10.1136/gutjnl-2014-308411. Epub 2015 Mar 9. PMID 25753029
- [Background] Sano Y, Tanaka S, Kudo SE, Saito S, Matsuda T, Wada Y, Fujii T, Ikematsu H, Uraoka T, Kobayashi N, Nakamura H, Hotta K, Horimatsu T, Sakamoto N, Fu KI, Tsuruta O, Kawano H, Kashida H, Takeuchi Y, Machida H, Kusaka T, Yoshida N, Hirata I, Terai T, Yamano HO, Kaneko K, Nakajima T, Sakamoto T, Yamaguchi Y, Tamai N, Nakano N, Hayashi N, Oka S, Iwatate M, Ishikawa H, Murakami Y, Yoshida S, Saito Y. Narrow-band imaging (NBI) magnifying endoscopic classification of colorectal tumors proposed by the Japan NBI Expert Team. Dig Endosc. 2016 Jul;28(5):526-33. doi: 10.1111/den.12644. Epub 2016 Apr 20. PMID 26927367
- [Background] Hewett DG, Kaltenbach T, Sano Y, Tanaka S, Saunders BP, Ponchon T, Soetikno R, Rex DK. Validation of a simple classification system for endoscopic diagnosis of small colorectal polyps using narrow-band imaging. Gastroenterology. 2012 Sep;143(3):599-607.e1. doi: 10.1053/j.gastro.2012.05.006. Epub 2012 May 15. PMID 22609383
- [Background] Dixon MF. Gastrointestinal epithelial neoplasia: Vienna revisited. Gut. 2002 Jul;51(1):130-1. doi: 10.1136/gut.51.1.130. PMID 12077106
- [Background] Nagtegaal ID, Odze RD, Klimstra D, Paradis V, Rugge M, Schirmacher P, Washington KM, Carneiro F, Cree IA; WHO Classification of Tumours Editorial Board. The 2019 WHO classification of tumours of the digestive system. Histopathology. 2020 Jan;76(2):182-188. doi: 10.1111/his.13975. Epub 2019 Nov 13. No abstract available. PMID 31433515
- [Derived] Ortiz O, Daca-Alvarez M, Rivero-Sanchez L, Gimeno-Garcia AZ, Carrillo-Palau M, Alvarez V, Ledo-Rodriguez A, Ricciardiello L, Pierantoni C, Huneburg R, Nattermann J, Bisschops R, Tejpar S, Huerta A, Riu Pons F, Alvarez-Urturi C, Lopez-Vicente J, Repici A, Hassan C, Cid L, Cavestro GM, Romero-Mascarell C, Gordillo J, Puig I, Herraiz M, Betes M, Herrero J, Jover R, Balaguer F, Pellise M; TIMELY study group. An artificial intelligence-assisted system versus white light endoscopy alone for adenoma detection in individuals with Lynch syndrome (TIMELY): an international, multicentre, randomised controlled trial. Lancet Gastroenterol Hepatol. 2024 Sep;9(9):802-810. doi: 10.1016/S2468-1253(24)00187-0. Epub 2024 Jul 19. PMID 39033774